CLINICAL TRIAL: NCT04822285
Title: Psychological Triaging Intervention: Rescue From Psychological Distress and Improving Senior Nursing Students' Resilience Capacity During COVID-19 Crisis
Brief Title: Effect Psychological Triaging Intervention on Students' Psychological Distress and Resilience Capacity
Acronym: Triaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Rasha salah elsayed eweida, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1522112020
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Psychological Distress; Resilience
Keywords: Psychological Distress; Triage; Resilience; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychological Triaging Intervention (Experimental): The PTI intervention followed the path of RAPID Psychological First Aid model of John Hopkins University (Everly& Lating 2012). The content of the PTI represents a simple structure that is revolved around five core phases including (R: establishing rapport and reflective listening, A: assessment, P: prioritization, I: intervention and D: disposition& follow up).
  Interventions: Behavioral: Psychological Triaging Intervention
- Routine Psychological support (Active Comparator): For the comparison group, the researchers provided them with routine psychological support that mainly revolved around enhancing their self-compassion, practicing mindfulness exercises, keeping them socially connected with their family and peers. Moreover, adopt a healthy lifestyle such as; engage in physical activity, eating a well-balanced diet, and sleeping well.
  Interventions: Behavioral: Routine psychological support

INTERVENTIONS:
Behavioral: Psychological Triaging Intervention — The PTI intervention followed the path of RAPID Psychological First Aid model of John Hopkins University (Everly& Lating 2012). The content of the PTI represents a simple structure that is revolved around five core phases including (R: establishing rapport and reflective listening, A: assessment, P: prioritization, I: intervention and D: disposition& follow up).
  Arms: Psychological Triaging Intervention
Behavioral: Routine psychological support — For the comparison group, the researchers provided them with routine psychological support that mainly revolved around enhancing their self-compassion, practicing mindfulness exercises, keeping them socially connected with their family and peers. Moreover, adopt a healthy lifestyle such as; engage in physical activity, eating a well-balanced diet, and sleeping well.
  Arms: Routine Psychological support

SUMMARY:
This study aimed to investigate the effect of the psychological triaging intervention (PTI) on the psychological distress and resilience capacity levels among the intern-nursing students during the COVID-19 crisis.

Research Hypothesis

Intern-nursing students who attend PTI exhibit lower COVID-19 related psychological distress level and higher resilience capacity than those who receive routine psychological support.

DETAILED DESCRIPTION:
The intern-nursing students' psychological well-being and resilience are of indispensable significance during these unprecedented days. 64 Intern-nursing students. Sixty-four intern-nursing students who completed a preliminary survey and demonstrated both high level of psychological distress and low resilience capacity as a result of their exposure to patients with COVID-19 during their internship period were randomly assigned to two equal groups and the study group were engaged in the PTI intervention which followed the path of RAPID Psychological First Aid model.

The PTI intervention followed the path of RAPID Psychological First Aid model of John Hopkins University (Everly& Lating 2012). The content of the PTI represents a simple structure that is revolved around five core phases including (R: establishing rapport and reflective listening, A: assessment, P: prioritization, I: intervention and D: disposition& follow up).

ELIGIBILITY:
Inclusion Criteria:

* Exposed to patients with COVID-19

Exclusion Criteria:

* Did not exposed to patients with COVID-19

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2021-03-21 (Actual)

PRIMARY OUTCOMES:
severity of psychological distress | " 2 weeks "
  The General Health Questionnaire (GHQ-12) was developed by (Goldberg, 1972). The questionnaire comprises 12- self-report items to measure the severity of psychological distress. The presence the symptoms was rated on 4- points Likert-type scale; (0="not at all present", 1="same as usual present"; 2="rather more than usual present"; 3="much more than usual present"). The tool demonstrated high reliability as Cronbach's alpha coefficient was 0.87. The total score ranged from 0-36. The higher score representing higher level of psychological distress.

OTHER OUTCOMES:
Resilience Capacity | " 2 weeks "
  It consists of 25-item to assess the resilience capacity. The CD-RISC was abridged to 10 items to reflect the individuals' ability to tolerate painful experience. Such as; ability to adapt to change, tendency to bounce back after hardship and ability to stay focused under pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Eman m Taha, professor, Study Chair — Alexandria University
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bozdag F, Ergun N. Psychological Resilience of Healthcare Professionals During COVID-19 Pandemic. Psychol Rep. 2021 Dec;124(6):2567-2586. doi: 10.1177/0033294120965477. Epub 2020 Oct 13. PMID 33050800
- [Background] Eweida RS, Rashwan ZI, Desoky GM, Khonji LM. Mental strain and changes in psychological health hub among intern-nursing students at pediatric and medical-surgical units amid ambience of COVID-19 pandemic: A comprehensive survey. Nurse Educ Pract. 2020 Nov;49:102915. doi: 10.1016/j.nepr.2020.102915. Epub 2020 Nov 10. PMID 33227694
- [Background] Farkas D, Orosz G. Ego-resiliency reloaded: a three-component model of general resiliency. PLoS One. 2015 Mar 27;10(3):e0120883. doi: 10.1371/journal.pone.0120883. eCollection 2015. PMID 25815881
- [Background] Maben J, Bridges J. Covid-19: Supporting nurses' psychological and mental health. J Clin Nurs. 2020 Aug;29(15-16):2742-2750. doi: 10.1111/jocn.15307. Epub 2020 Jun 2. No abstract available. PMID 32320509
- [Background] Prime H, Wade M, Browne DT. Risk and resilience in family well-being during the COVID-19 pandemic. Am Psychol. 2020 Jul-Aug;75(5):631-643. doi: 10.1037/amp0000660. Epub 2020 May 21. PMID 32437181
- [Background] Shultz JM, Forbes D. Psychological First Aid: Rapid proliferation and the search for evidence. Disaster Health. 2013 Aug 2;2(1):3-12. doi: 10.4161/dish.26006. eCollection 2014 Jan-Mar. PMID 28228996